CLINICAL TRIAL: NCT02860598
Title: Clinical Observatory of the Prescription of Erythropoietin as Treatment of Anemia Induced by Chemotherapy or Allograft Conditioning Among the Patients With a Haematological Malignancy
Brief Title: Observatory of the Prescription of Erythropoietin as Treatment of Anemia Induced by Chemotherapy or Allograft Conditioning Among the Patients With a Haematological Malignancy
Acronym: EPREX/LAM-ALLO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0419
Record Dates: First submitted 2016-07-20; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-06

CONDITIONS: Anemia; Acute Myeloid Leukemia
Keywords: ESAs; erythropoietin; AML; HSCT
MeSH Terms: conditions — Anemia; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Patient with AML de novo or secondary myelodysplasia, in Complete Remission (CR) after induction and / or salvage therapy and candidate to receive a consolidation therapy
- Group 2: Patient with hematologic malignancies (ALL, AML, chronic lymphocytic leukemia (CLL), non-Hodgkin lymphoma, myeloma, myeloproliferative syndrome (MDS)) and candidate for blood marrow or stem cell or placental blood transplantation.

SUMMARY:
Anemia concerns a lot of patients with cancer and affects their quality of life (QOL). Numerous studies in oncology have demonstrated the benefit of erythropoiesis-stimulating agents (ESA) in the treatment of anemia. ESAs allow the improvement of QOL,of the hemoglobin level (Hb) and is a validated alternative to transfusion.

However, in hematology, if there are some specific recommendations for the use of ESAs in lymphoid pathology, there are none for myeloid disorders and in the context of autografts and allogeneic hematopoietic stem-cell transplantation (HSCT). Thus, the investigators are in particular interested in both indications: treatment of anemia in acute myeloid leukemia (AML) patients treated with chemotherapy, and the in patients receiving a myeloablative or a non-myeloablative conditioning before allogeneic HSCT, whatever type of donor and cell source.

DETAILED DESCRIPTION:
In this context, a prospective observatory was conducted from 2006 to 2009 in the hematology department of Prof. Michallet to assess the impact of prescribing ESAs (epoetin beta and darbepoetin) for these two distinct patient populations. A significant improvement in QOL during the six-month follow- up was observed in both groups. The effectiveness of the ESA on the red cell recovery and the reduction of red blood cell transfusions was established by comparing the evolution of Hb and transfusion needs of the population under ESA to a matched population. Moreover, no significant difference in the occurrence of thromboembolic events in survival and progression-free survival was observed between the ESA group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patient with AML de novo or secondary myelodysplasia in Complete Remission (CR) after induction and / or salvage therapy and candidate to receive a consolidation therapy.
* OR Patient with hematologic malignancies (ALL, AML, chronic lymphocytic leukemia, CLL, non-Hodgkin lymphoma, MDS, myeloma, myeloproliferative syndrome) and candidate for blood marrow or stem cell or placental blood transplantation.

Depending on the hematologic malignancy, pre-transplant status of patients included will be the CR, very good partial or partial response.

* Patient with anemia (Hb blood level ≤ 110g / l) induced by consolidation chemotherapy or allograft conditioning (myeloablative or non-myeloablative).
* Patient eligible according to the investigator, to treatment with ESA (evaluation by the investigator of the benefice- risk ratio).
* Written informed consent.

Exclusion Criteria:

* Contraindication to epoetin alfa or epoetin zeta.
* Patient not able to receive adequate antithrombotic prophylaxis.
* Patients who received ESA therapy within 3 weeks prior to inclusion.
* non French-speaking patient
* Patient participating or having participated to a clinical trial evaluating a novel molecule in the 30 days before inclusion.
* pregnant or nursing, woman or woman of childbearing potential without effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with AML de novo or secondary myelodysplasia in Complete Remission (CR) after induction and / or salvage therapy and candidate to receive a consolidation therapy.
  OR Patient with hematologic malignancies (ALL, AML, chronic lymphocytic leukemia, CLL, non-Hodgkin lymphoma, MDS, myeloma, myeloproliferative syndrome) and candidate for blood marrow or stem cell or placental blood transplantation.
Sampling Method: Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2011-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Change in the Haemoglobin level from the inclusion to the final visit | At Day 1 and Month 6

SECONDARY OUTCOMES:
Change in Fact-An questionnaire score | At Day 1 and Month 6
  Patient's quality of life: Fact-An questionnaire
Change in Fact-An subscales | At Day 1 and Month 6
  Patient's quality of life: Fact-An subscales
Change in Fact-G questionnaire score | At Day 1 and Month 6
  Patient's quality of life: Fact-G questionnaire (including physical well-being, social well-being, emotional well-being and functional well-being)
Change in Fact-Anemia questionnaire score | At Day 1 and Month 6
  Patient's quality of life: Fact-Anemia (including Fact-Fatigue)
Change in the Number of red blood cell transfusions | At Month 3 and Month 6
  Data on the erythrocyte recovery
Change in the Number of platelet transfusions | At Month 3 and Month 6
  Data on the platelet recovery

CONTACTS AND LOCATIONS:
Overall Officials: Mauricette Michallet, Prof., Study Director — Hematology Department, Hospices Civils de Lyon
Locations (1):
- Jeremy MONFRAY, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No